CLINICAL TRIAL: NCT05727267
Title: TherVacB_Phase1a: Open Phase 1a Trial to Assess the Safety and Immunogenicity of a Heterologous Protein Prime/MVA Boost Therapeutic Hepatitis B Vaccine Candidate in Healthy Volunteers
Brief Title: A Heterologous Protein Prime/MVA Boost Therapeutic Hepatitis B Vaccine Candidate
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Center for Infection Research (Other); Medical Biometry and Epidemiology_- Universitätsklinikum Hamburg Eppendorf (Unknown); Helmholtz Zentrum München (Industry); The Fraunhofer-Gesellschaft (Other); Institute of Virology Helmholtz Zentrum München (HMGU) (Unknown); LMU Klinikum (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TherVacB_Phase1
Record Dates: First submitted 2022-11-06; First posted 2023-02-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Heplisav-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm A0 (Experimental): HEPLISAV B® and MVA-HBVac high dose
  Interventions: Biological: HEPLISAV B; TherVacB
- Arm B0.1 (Experimental): HEPLISAV B® & HBcoreAg low dose and MVA-HBVac low dose
  Interventions: Biological: HEPLISAV B; TherVacB
- Arm B0.2 (Experimental): 2 x HEPLISAV B® & HBcoreAg medium and MVA-HBVac high dose
  Interventions: Biological: HEPLISAV B; TherVacB
- Arm C0.1 (Experimental): HBsAg high dose & HBcoreAg high dose and MVA-HBVac high dose
  Interventions: Biological: TherVacB
- Arm C0.2 (Experimental): HBsAg medium dose + adjuvant low dose & HBcoreAg medium dose and MVA-HBVac high dose
  Interventions: Biological: TherVacB
- Arm C0.3 (Experimental): HBsAg high dose + adjuvant & HBcoreAg high dose and MVA-HBVac high dose
  Interventions: Biological: TherVacB

INTERVENTIONS:
Biological: HEPLISAV B; TherVacB — Administration of the described combinations via the intramuscular route
  Arms: Arm A0; Arm B0.1; Arm B0.2
Biological: TherVacB — Administration of the described combinations via the intramuscular route
  Arms: Arm C0.1; Arm C0.2; Arm C0.3

SUMMARY:
This study is an open-label, ascending dose phase 1a trial to assess the safety and immunogenicity of a heterologous protein prime/MVA boost therapeutic hepatitis B vaccine

DETAILED DESCRIPTION:
The clinical trial is divided into two overlapping parts (part I and part II) in 24 healthy male and female subjects aged 18-65 years.

Part I (N = 11) Protein prime vaccinations two times (day 0 and 28) and MVA based boost vaccination 1 x (day 56) 3 subjects will be allocated to A0 and receive HEPLISAV B® and a boost with MVA-HBVac high dose 3 subjects will be allocated to B0.1 and receive HEPLISAV B® & HBcoreAg low dose and a boost with MVA-HBVac low dose 5 subjects will be allocated to B0.2 and receive 2 x HEPLISAV B® & HBcoreAg medium dose and a boost with MVA-HBVac high dose Part II (N = 13) Protein prime vaccinations two times (day 0 and 28) and MVA based boost with MVA-HBVac high dose on day 56 3 subjects will be allocated to C0.1 and receive HBsAg high dose & HBcoreAg high dose plus boost 5 subjects will be allocated to C0.2 and receive HBsAg medium dose + adjuvant low dose & HBcoreAg medium dose plus boost 5 subjects will be allocated to C0.3 and receive HBsAg high dose + adjuvant &HBcoreAg high dose plus boost

ELIGIBILITY:
Key inclusion criteria:

1. Ability to understand the subject information and to personally name, sign and date the informed consent to participate in the clinical trial.
2. Provided written informed consent.
3. Healthy male and female subjects aged 18-65 years at time of informed consent.
4. No clinically significant health problems as determined during medical history and physical examination and clinical laboratory results at screening visit. The following laboratory parameters should be within normal limits: WBC, ANC, platelets. AST and ALT should be ≤ULN, CrCL >60mL/min and total bilirubin should not exceed 1,5 x ULN. Non-clinically significant, minor deviations of laboratory measurements can be tolerated as they will not increase the risk of the individual having an adverse outcome from participating in this clinical trial as judged by the investigator.
5. Participant may be on chronic or as needed medications if, in the opinion of the investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity and do not indicate worsening of a pre-existing medical condition.
6. Body mass index 18.5-32.0 kg/m2 and weight >50 kg at screening.
7. Women of child-bearing potential (WOCBP) only: non-pregnant, non-lactating women with negative pregnancy test.
8. WOCBP who agree to comply with the applicable contraceptive requirements of the protocol.

Key exclusion criteria:

1. Receipt of any vaccine in the 2 weeks prior to first trial vaccination (4 weeks for live vaccines), or planned receipt of any vaccine in the 2 weeks before each trial vaccination (4 weeks for live vaccines) until 3 weeks following each trial vaccination. Exception: Required recommended pandemic and influenza vaccines are allowed.
2. Previous hepatitis B vaccination or an anti-HBs positive serum status before study start.
3. Immunization with a poxvirus-based viral vector. A suspected or confirmed monkeypox infection within the last 10 years.
4. Known allergy to components of the vaccine products (incl. hypersensitivity to yeast) or history of life-threatening reactions to vaccines containing one of the substances.
5. Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccines.
6. History of previous HBV infection (if serostatus: anti-HBc positive).
7. Clinically relevant findings in ECG or significant thromboembolic events in medical history.
8. Evidence for a condition in the subject's medical history or during medical examination that might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of vaccine pro-ducts.
9. Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years.
10. Any chronic or active neurologic disorder, including seizures, and epilepsy, excluding a febrile seizure as a child and occasional migraine headaches.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
occurence of solicited local reactogenicity signs and symptoms (AEs) | up to day 63
  numerbers of solicited AEs for 7 days after each vaccination
occurence of unsolicited local reactogenicity signs and symptoms | up to day 84
  numbers of of unsolicited AEs for 28 days after each vaccination
changes of safety laboratory measures | up to day 224
  changes of values from safety laboratory measures from baseline
nature, frequency and severity of adverse events associated with the vaccine | up to day 224
  numbers and severity grade of SAEs throughout the period of the clinical trial

SECONDARY OUTCOMES:
Magnitude of anti-HBs antibody responses | day 0,day 7,day 28,day 35,day 56,day 63,day 70,day 84,day 224
  determined by an accredited serological immuno-assay
Percentage of participants who seroconvert to anti-HBs (>10 IU/l), anti-HBc or anti-HBs and anti-HBc | day 0,day 7,day 28,day 35,day 56,day 63,day 70,day 84,day 224
  determined by an accredited serological immuno-assay
Magnitude of HBV-specific T-cell responses | day 0,day 7,day 28,day 35,day 56,day 63,day 70,day 84,day 224
  determined by cytokine release assays

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M Addo, Prof, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Bernhard Nocht Centre for Clinical Trials (BNCCT), Hamburg
  - Division of Infectious Diseases and Tropical Medicine, LMU Klinikum, Munich

IPD SHARING:
Plan to Share IPD: No